CLINICAL TRIAL: NCT06151158
Title: Preventing Suicidal Behavior With Diverse High-Risk Youth in Acute Care Settings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Johns Hopkins All Children's Hospital (Other); Children's Hospital of Philadelphia (Other); Reichman University (Other); Patient-Centered Outcomes Research Institute (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00408733
Record Dates: First submitted 2023-11-21; First posted 2023-11-30 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Suicide, Attempted; Suicide Ideation; Suicide; Suicide Prevention
Keywords: Safety Planning Intervention; Ultra-Brief Crisis; Interpersonal Psychotherapy for Adolescents; Emergency Department; Suicide Prevention
MeSH Terms: conditions — Suicide, Attempted; Suicide; Suicide Prevention; Emergencies | interventions — Interpersonal Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Safety Planning Intervention (Active Comparator): The SPI is a brief, evidence- based intervention that provides people with an individualized set of steps that can be used progressively to both reduce risk and maintain safety when suicide ideation (SI) emerges. Safety plans are developed collaboratively between providers, at risk youth, and family members when possible. Core SPI components include recognizing warning signs of an imminent suicidal crisis (e.g., changes in mood, thoughts or behaviors); using internal coping skills to reduce distress; using people or places in the individual's support network as a means of distraction from SI; reaching out to family or friends to help manage the crisis; contacting health professionals or emergency services; and reducing access to lethal means. SPI+ includes a brief follow-up component post- discharge that includes contacting the patient for a mood and risk check-in; reviewing and revising the safety plan; and facilitating connection with community mental health services.
  Interventions: Behavioral: Stanley Brown Safety Planning Intervention and Follow-up Contacts (SPI+)
- Ultra-Brief Crisis IPT-A (Active Comparator): Interpersonal Psychotherapy for Adolescents Ultra Short Crisis Intervention (IPT-A SCI) is a scalable, flexible, and extensively examined mental health treatment developed to reduce depressive symptoms and improve interpersonal functioning, and has been adapted for use in adolescents (IPT-A SCI) and shown to be effective in treating depression and reducing associated suicide risk. Interpersonal problems are often at the core of suicidal thinking and behavior in youths including minority youths.
  Interventions: Behavioral: Interpersonal Psychotherapy for Adolescents Ultra Short Crisis Intervention (IPT-A SCI)

INTERVENTIONS:
Behavioral: Stanley Brown Safety Planning Intervention and Follow-up Contacts (SPI+) — Stanley Brown Safety Planning completed in the emergency department with 3 follow-up contacts after discharge
  Arms: Safety Planning Intervention
Behavioral: Interpersonal Psychotherapy for Adolescents Ultra Short Crisis Intervention (IPT-A SCI) — Five session crisis focused version of IPT for adolescents.
  Arms: Ultra-Brief Crisis IPT-A

SUMMARY:
The study will compare the effectiveness of two relatively brief and scalable evidence-based interventions: the Stanley Brown Safety Planning Intervention and Follow-up Contacts (SPI+), a suicide-specific intervention that helps people prevent suicidal crises from escalating, and Interpersonal Psychotherapy for Adolescents Ultra Short Crisis Intervention (IPT-A SCI), a psychotherapeutic crisis intervention treatment for suicidal adolescents that teaches youth skills to prevent suicidal crises and addresses interpersonal problems that lead to suicidal crises. The results will inform the future standard of care for youth at risk for suicide presenting in the ED setting. This project focuses on suicidal youth ages 12-19 in three ethnically and racially diverse urban areas: Philadelphia, Pennsylvania; Baltimore, Maryland; and upper Manhattan/lower Bronx in New York City.

DETAILED DESCRIPTION:
Emergency department (ED) visits for suicide-related concerns have been increasing in youth over the past decade, a trend potentially exacerbated by the COVID-19 pandemic. Also, youth suicidal thoughts and attempts have increased with the 2019 Centers for Disease Control and Prevention (CDC) Youth Risk Behavior Surveillance System (YRBSS) finding that 18.8 percent of high school students have seriously considered suicide and 8.9 percent had attempted suicide in the past year. Furthermore, suicide rates are increasing more rapidly in Latino/Latina, Black, and multiracial youth, especially Black youth as compared to White youth. Similar increases in suicide risk are seen in lesbian, gay, bisexual, transgender, queer and other sexually minority (LGBTQ+) youth. This project focuses on suicidal youth ages 12-19 in three ethnically and racially diverse urban areas: Philadelphia, Pennsylvania; Baltimore, Maryland; and upper Manhattan/lower Bronx in New York City.

There is limited evidence about which interventions are most helpful for suicidal youth in acute care settings such as EDs. Interventions like safety planning (Safety Planning Intervention with follow-up contacts) are delivered primarily in ED settings while others like Interpersonal Psychotherapy for Adolescents Ultra Short Crisis Intervention (IPT-A SCI) are provided primarily in outpatient settings. Furthermore, safety planning focuses on deescalating suicidal crises when beginning to occur, while IPT-A SCI focuses on developing skills to prevent crises from occurring. While both approaches have an evidence base, it is not yet known which one is more effective and acceptable in a diverse youth population. Determining which intervention is more effective has implications for dissemination and resource allocation to EDs or outpatient settings.

The research team includes a group of ethnically and racially diverse partners and advisors, advocates, researchers, ED physicians, nurses, and social workers, some of whom have lived experience of suicide attempts and suicide loss. This team has provided feedback about crucial elements of this proposal, e.g., recruitment, intervention approaches, and follow-up approaches and will continue active involvement in all stages of this project.

The study will compare the effectiveness of two relatively brief and scalable evidence-based interventions: the SPI+, a suicide-specific intervention that helps people prevent suicidal crises from escalating, and IPT-A SCI, a psychotherapeutic crisis intervention treatment for suicidal adolescents that teaches youth skills to prevent suicidal crises and addresses interpersonal problems that lead to suicidal crises. The results will inform the future standard of care for youth at risk for suicide presenting in the ED setting.

ELIGIBILITY:
Inclusion Criteria:

* Acute care visit for suicide-related concern or screen positive on a suicide risk screener (serious SI as indicated by a C-SSRS screening endorsing question two "Have you actually had any thoughts of killing yourself?" in past four weeks or SA in past four weeks);
* Has a cell phone with ability to receive phone calls and text messages over the 12-month follow-up;
* Ability to speak, understand, and read in English or Spanish

Exclusion Criteria:

* Significant cognitive or developmental delays that prevent understanding or using SPI or IPT-A SCI. Participants must be verbally fluent and have the ability to communicate verbally. This will, in part, be determined by notes in Epic and/or by asking one of the patient's parents/clinicians;
* Altered mental status that precludes ability to provide informed assent or consent (acute psychosis, intoxication, or mania);
* Unable to provide informed consent (adults); assent (minors); permission (parents/caregivers).

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2028-10-14 (Estimated); Study Completion 2028-10-14 (Estimated)

PRIMARY OUTCOMES:
Change in Suicidal ideation as assessed by the Suicide Assessment Five-step Evaluation and Triage (SAFE-T) with Columbia-Suicide Severity Rating Scale (C-SSRS) Recent | baseline, 3 months, 6 months, 12 months
  Suicidal thoughts: measured using the Suicide Assessment Five-step Evaluation and Triage (SAFE-T) with Columbia-Suicide Severity Rating Scale (C-SSRS) Recent. Scores for suicidal ideation range from 0 to 5, with higher scores indicating more serious suicidal ideation, where 0 = "no suicidal thoughts"; 1= "wish to be dead"; 2 = "nonspecific active suicidal thoughts"; 3 = "suicidal thoughts with methods"; 4 = "suicidal intent"; and 5 = "suicidal intent with plan".
Change in Suicidal behavior as assessed by the Suicide Assessment Five-step Evaluation and Triage (SAFE-T) with Columbia-Suicide Severity Rating Scale (C-SSRS) Recent | baseline, 3 months, 6 months, 12 months
  Suicidal behavior with intent to die: measured using the Suicide Assessment Five-step Evaluation and Triage (SAFE-T) with Columbia-Suicide Severity Rating Scale (C-SSRS) Recent. Scored 0 to 1, with 1 indicating a suicide attempt since last assessment.
Number of Suicides | 12 months
  Measured through Death Records or Suicide from Office of Chief Medical Examiner, family report or medical record

SECONDARY OUTCOMES:
Change in Frequency of mental health service utilization as assessed by Services Assessment for Children and Adolescents (SACA) | baseline, 3 months, 6 months, 12 months
  Services Assessment for Children and Adolescents (SACA) use of inpatient, outpatient, school services since last assessment. Items are dichotomous (yes/no) and the scale ranges from 0 (no services) to 3 (3 types of services), higher numbers indicate more services.
Change in Self reported Quality of Life as assessed by the Euro-Qol 5-Dimension 3-level tool (EQ-5D-3L) | baseline, 3 months, 6 months, 12 months
  Euro-Qol 5-Dimension 3-level tool (EQ-5D-3L) for young adults. The scale consists of a descriptive system that comprises five items referring to the domains mobility, self-care, usual activities, pain/discomfort and anxiety/depression scored as presenting no problems, moderate problems or severe problems. Each of the five items (range 0-2) with higher scores indicating better quality of life. A component of this scale is the EuroQol visual analogue scale (EQ-VAS) which participants can use a number from 0 (the worst) -100 (the best health state imaginable).
Change in Self reported Quality of Life as assessed by the Euro-Qol 5-Dimension Youth (EQ-5D-Y) | baseline, 3 months, 6 months, 12 months
  Quality of Life will be assessed by the Euro-Qol 5-Dimension Youth (EQ-5D-Y). The scale consists of a descriptive system that comprises five items referring to the domains mobility, self-care, usual activities, pain/discomfort and anxiety/depression scored as presenting no problems, moderate problems or severe problems. Each of the five items (range 0-2) with higher scores indicating better quality of life. A component of this scale is the EuroQol visual analogue scale (EQ-VAS) which participants can use a number from 0 (the worst) -100 (the best health state imaginable).
Change in Generalized Anxiety Disorder as assessed by the The Generalized Anxiety Disorder 7 question scale (GAD-7). | baseline, 3 months, 6 months, 12 months
  Generalized Anxiety Disorder will be assessed by the GAD 7 question scale. The Generalized Anxiety Disorder 7 is a self-reported questionnaire for screening and severity measuring of generalized anxiety disorder. The GAD-7 total score ranges from 0 to 21 with clinical categorizations of anxiety levels as follows: GAD-7 score of 0-4 (none), 5-9 (mild), 10-14 (moderate), and 15-21 (severe).
Change in Depression severity as assessed by the nine-item Patient Health Questionnaire (PHQ-9). | baseline, 3 months, 6 months, 12 months
  The nine-item Patient Health Questionnaire is a depressive symptom scale and diagnostic tool that assesses the presence and severity of depressive symptoms and a possible depressive disorder. The PHQ-9 total score ranges from 0 to 27 (scores of 5-9 are classified as mild depression; 10-14 as moderate depression; 15-19 as moderately severe depression; ≥ 20 as severe depression).
Change in conflicts with family members as assessed by the Conflict Behavior Questionnaire (CBQ). | baseline, 3 months, 6 months, 12 months
  The Conflict Behavior Questionnaire (CBQ) reliably assesses the adolescent's perception of their relationship with their parents. The CBQ total score ranges from 0-20, with higher scores indicating greater conflict with each parent.
Change in social interactions with peers as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Peer Relationships scale. | baseline, 3 months, 6 months, 12 months
  The PROMIS (Patient-Reported Outcomes Measurement Information System) scale assesses social interactions with peers. The Pediatric Peer Relationships scale has a possible score between 1 and 40, with higher scores indicating greater social interactions with peers.
Change in social interactions with family as assessed by the Patient-Reported Outcomes Measurement Information System (PROMIS) Pediatric Family Relationships scale. | baseline, 3 months, 6 months, 12 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) scale assesses social interactions with family. The Pediatric Family Relationships scale has a possible score between 1 and 40, with higher scores indicating greater social interactions with family.
Change in skill use derived from the Stanley Brown Safety Planning Intervention and Follow-up Contacts (SPI+) arm | 3 months, 6 months, 12 months
  Project-created a self-report of Stanley Brown Safety Planning Intervention and Follow-up Contacts (SPI+) skill use during follow-up, indicating feasibility/acceptability of SPI, helpfulness of different skills/sections of the safety plan, and frequency of use for different skills/sections of the safety plan.
Change in skill use derived from the Interpersonal Psychotherapy for Adolescents Ultra Short Crisis Intervention (IPT-A SCI) arm | 3 months, 6 months, 12 months
  Project created a self-report of Interpersonal Psychotherapy for Adolescents Ultra Short Crisis Intervention (IPT-A SCI) skill use during follow-up indicating which components adolescents have used. The self-report survey scoring will be a summation and then taking an average of the sum to be the score. Higher scores closer to 5 indicate adolescents learned a lot of from the intervention, and the lower scores indicate adolescents learned few skills.

CONTACTS AND LOCATIONS:
Overall Officials: Holly C Wilcox, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (6):
- United States (6):
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Johns Hopkins University, Baltimore, Maryland
  - Columbia University Irving Medical Center (CUMC), New York, New York
  - Weill-Cornell Medicine, New York, New York
  - University of North Carolina Medical Center, Chapel Hill, North Carolina
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stanley B, Brown GK, Brenner LA, Galfalvy HC, Currier GW, Knox KL, Chaudhury SR, Bush AL, Green KL. Comparison of the Safety Planning Intervention With Follow-up vs Usual Care of Suicidal Patients Treated in the Emergency Department. JAMA Psychiatry. 2018 Sep 1;75(9):894-900. doi: 10.1001/jamapsychiatry.2018.1776. PMID 29998307
- [Result] Haruvi Catalan L, Levis Frenk M, Adini Spigelman E, Engelberg Y, Barzilay S, Mufson L, Apter A, Benaroya Milshtein N, Fennig S, Klomek AB. Ultra-Brief Crisis IPT-A Based Intervention for Suicidal Children and Adolescents (IPT-A-SCI) Pilot Study Results. Front Psychiatry. 2020 Dec 9;11:553422. doi: 10.3389/fpsyt.2020.553422. eCollection 2020. PMID 33362595
- See also: Patient-Centered Outcomes Research Institute (PCORI) website description of study — https://www.pcori.org/research-results/2022/preventing-suicidal-behavior-diverse-high-risk-youth-acute-care-settings